CLINICAL TRIAL: NCT04521075
Title: A Phase Ib Trial to Evaluate the Safety and Efficacy of Fecal Microbial Transplantation (FMT) in Combination With Nivolumab in Subjects With Metastatic or Inoperable Melanoma, Microsatellite Instability-high (MSI-H) or Mismatch-repair Deficient (dMMR) Cancer, or Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Phase Ib Trial to Evaluate the Safety and Efficacy of FMT and Nivolumab in Subjects With Metastatic or Inoperable Melanoma, MSI-H, dMMR or NSCLC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ella Therapeutics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6735-19
Record Dates: First submitted 2020-08-13; First posted 2020-08-20 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Melanoma Stage IV; Unresectable Melanoma; NSCLC Stage IV
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: Stage I:
  Cohort A: Fifteen Melanoma patients will be treated with FMT capsules originating from 5 different donors.
  Cohort B: Two NSCLC patients will be treated with FMT capsules originating from 2 different donors.
  Cohort C: Three MSI-H or dMMR patients will be treated with FMT via colonoscopy and capsules combined with anti-PD-1 (Nivolumab).
  An interim analysis will be conducted following completion of recruitment of 15 patients.
  Based on the interim analysis, the abovementioned independent cohorts will be expanded to include additional patients as
  Stage II:
  Cohort A expansion will include 15 melanoma patients Cohort C expansion will include seven MSI-H or dMMR patients.
  Patients will be treated with FMT originating from selected donors, combined with anti-PD-1 (Nivolumab).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental): Combination treatment: anti PD1 + FMT by capsules
  Interventions: Biological: Fecal Microbial Transplantation by capsules

INTERVENTIONS:
Biological: Fecal Microbial Transplantation by capsules — Cohorts A and B - Patients will receive 30 oral capsules per administration for two consecutive days (Days 1-2) Cohort C - Patients will receive FMT via colonscopy (Day 1), followed the day after by adnistration of 12 oral capsules (Day 2)
  Combination cycles: 6 combined cycles Q2W of FMT maintenance followed by treatment with anti-PD1. Anti-PD-1 will be administered at least one day and up to 3 days after the FMT.
  Maintenance of FMT by oral capsules: 12 capsules per administration. Anti PD-1 therapy: A dose of 240 mg Nivolumab will be administrated by intravenous infusion.
  Other Names: Nivolumab

SUMMARY:
A Phase Ib trial to evaluate the safety and efficacy of Fecal Microbial Transplantation (FMT) in combination with Nivolumab in subjects with metastatic or inoperable melanoma, microsatellite instability-high (MSI-H) or mismatch-repair deficient (dMMR) cancer, or Non-Small Cell Lung Cancer (NSCLC)

DETAILED DESCRIPTION:
This study is a Phase I single-center adaptive design study to evaluate the safety and efficacy of FMT in combination with Nivolumab for adult subjects with treatment-refractory or inoperable melanoma, MSH-H, dMMr or NSCLC.

FMT will be conducted with fecal capsules, originating from patients that have achieved a durable complete response with immune checkpoint inhibitors. The study will evaluate the safety and efficacy of the combination of FMT with Nivolumab, a human immunoglobulin G4 (IgG4) monoclonal antibody that blocks PD-1 (anti PD-1) treatment and explore different biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Age and gender: 18 and older, all genders
2. Signed written informed consent . Participants must be willing to participate in the study and provide written and signed informed consent (ICF) for the study.

   Participants must be willing and able to complete all study specific procedures and visits
3. Diagnosis:

   For NSCLC patients Histologically or cytologically confirmed metastatic or locally advanced non-small cell lung cancer not amenable to curative treatment that have a confirmed progression on anti-PD-1/PDL1 therapy:

   Subjects may have had a maximum of one prior line of therapy after failure of anti-PD-1/ Programmed death-ligand 1 (PDL1) therapy Received a platinum based chemotherapy for non-small cell lung cancer; or, Subjects with a documented activating mutation {e.g., against epidermal growth factor receptor (EGFR), against rearranged anaplastic lymphoma kinase (ALK), Proto-oncogene tyrosine-protein kinase (ROS)} must have received the appropriate targeted therapy.

   For Melanoma patients Histologically confirmed unresectable or metastatic melanoma not amenable to curative treatment that have a confirmed progression on anti-PD-1/PD-L1 therapy: a. Subjects may have had a maximum of one prior line of therapy after failure of anti-PD-1/PDL1 therapy b. Subjects with a documented B-Raf (BRAF) mutation must have received the appropriate targeted therapy

   For MSI-H/dMMR patients -Histologically confirmed MSI-H/dMMR metastatic solid tumors including the following indications: colorectal adenocarcinoma, gastric adenocarcinoma, esophageal adenocarcinoma, endometrial carcinoma, ovarian carcinoma, pancreatic ductal adenocarcinoma and urothelial carcinoma that had a confirmed progression on anti-PD-1/PD-L1-based therapy.
4. Biopsies Patients must agree to study biopsies at two time points: a. Pretreatment and on treatment gut biopsies. b. Pretreatment and on treatment tumor biopsies.
5. Measurable disease by RECIST v1.1.
6. Patient status: a. Eastern Cooperative Oncology Group (ECOG) status of 0-1 b. Liver function: Total bilirubin ≤ 2 Upper limit of normal (ULN), Alanine aminotransferase (ALT), and Aspartate aminotransferase (AST) ≤ 2.5 ULN (or < 5 in case of present liver metastasis) c. Neutrophils ≥ 1,000/mm3, platelets ≥ 100,000/mm3, Hb>8 g/dL d. Serum creatinine ≤ 1.5 ULN e. International normalized ratio (INR), prothrombin time (PT), and activated partial thromboplastin time (aPTT) ≤1.5x ULN
7. Pregnancy a. Negative urine or serum pregnancy test within 72 hours prior to receiving first dose of study procedure in women of childbearing potential. b. Use of an effective contraceptive method throughout the entire treatment period and up to 6 months after the completion of treatment in both males and females of child bearing potential.

Exclusion Criteria:

1. Medical Conditions :

   1.1 History of chronic or active colitis 1.2. Tumor involvement of the esophagus, stomach, small intestine or colo-rectum. Note: not applicable for patients with MSI-H or dMMR colorectal , gastric or esophageal adenocarcinoma 1.3. Has a current active or a past known additional malignancy within the last 5 years.

   1.4. Has an active or a documented history of autoimmune disease that required treatment in the past 2 years.

   1.5. Known food allergy to eggs, nuts, peanuts 1.6. Known allergy to neomycin,vancomycin or metronidazole 1.7. Pregnant or breastfeeding women 1.8. Has known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies) 1.9 Has known history of or is positive for hepatitis B or Hepatitis C.
2. Prior/Concomitant Therapy and medical procedure 2.1 Has ongoing immune-related adverse effects from previous immunotherapy treatments that are of Grade ≥2, excluding endocrine adverse effects 2.2 Immunosuppressive chronic treatments. Patients treated with Prednisone ≤10mg per day may be included.

   2.3 Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) or any major episode of infection requiring treatment with i.v. antibiotics or hospitalization (relating to the completion of the course of antibiotics, except if for tumor fever) within 28 days prior to the start of Day 1 2.4 Medical condition that requires chronic treatment with antibiotics 2.5 Vaccination with live vaccines within 28 days prior to start of Cycle 1, Day 1.

   2.6 Has received major surgery (within 28 days prior to the start of Cycle 1, Day 1), other than for diagnosis. Patient must have recovered from all surgery-related toxicities.

   2.7 Patient has a known intolerance to anti-PD-L1 or anti-PD1.
3. Prior/Concurrent Clinical Study Experience 3.1 Participation in another clinical trial with anti-neoplastic intervention up to 14 days prior to study entry
4. Other Exclusions 4.1 Any other serious uncontrolled medical condition (including active bleeding or non-healing wound) 4.2 Has known psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of FMT-related Adverse Events | 3 years
  Number of patients with adverse events that emerged post FMT. The AE severity grading scale for the NCI-CTCAE (v5.0) will be used for assessing AE severity
Overall Response Rate (ORR) | 3 years
  Number of patients with objective responses divided by the total number of evaluable patients, according to imaging studies (RECIST 1.1) and iRECIST

SECONDARY OUTCOMES:
Changes in immune activation in the gut | 3 years
  Immune activation in gut is defined as a 20% or more increase in cluster of differentiation 68 (CD68) cell counts pre and post FMT
Changes in immune activation in the tumor | 3 years
  Changes in the relative abundance of different immune cell population (such as the proportion of cluster of differentiation 8 (CD8) and T cell in the tumor pre and post FMT
Progression-free survival (PFS) | 3 years
  Duration of progression free status evaluated according to imaging studies (RECIST 1.1) and iRECIST.
To assess Overall survival (OS) | 3 years
  The proportion of patients remaining alive from initiation of study treatment until completion of two year follow-up from End of Treatment (EOT)
To assess Duration of response (DoR) | 3 years
  Time from initial response to disease progression or death among patients who have experienced a Complete Response (CR) or Partial Response (PR) according to RECIST v1.1
Incidence of immune related toxicities induced by anti-PD-1 | 3 years
  Number and Grade of immune related Adverse events (irAE) reported that emerged post anti-PD1 treatment

CONTACTS AND LOCATIONS:
Overall Officials: Guy Ben-Betzalel, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel